CLINICAL TRIAL: NCT00160082
Title: Efficacy and Safety of Xepol (Human Immunoglobulin) in Subjects With Post-Polio Syndrome (PPS): A Randomized, Two-Arm, Parallel, Double-Blind, Multi-Centre, Placebo Controlled Study
Brief Title: Efficacy and Safety of Xepol (Human Immunoglobulin) in Subjects With Post-Polio Syndrome (PPS)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Calliditas Therapeutics AB (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: IvIG 1/00
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2007-04-03 (Estimated); Status verified 2005-09

CONDITIONS: Post Polio Syndrome, PPS
Keywords: Post Polio Syndrome; PPS; Poliomyelitis; Paralylic Polio; Late effects of polio; Late onset polio sequele; Xepol; IvIg; Intravenous Immunoglobuline
MeSH Terms: conditions — Postpoliomyelitis Syndrome; Popliteal Pterygium Syndrome; Poliomyelitis

INTERVENTIONS:
Drug: Xepol

SUMMARY:
The primary objective was to assess the effect of Xepol compared to placebo on physical health and on muscle strength in subjects with post-polio syndrome.The secondary objective was to assess the effect of Xepol compared to placebo on functional balance, activity patterns, pain, fatigue, sleep, vitality, muscular strength, pulmonary capacity, walking ability, balance and safety.

DETAILED DESCRIPTION:
Study Rationale:

In an earlier open and non-controlled study in 10 patients with PPS, Xepol was given during three days. The patients showed improvements in muscular strength and co-ordination and a decrease in pain. The aim of this study was to investigate if these findings can be confirmed in a larger, double-blind, randomised and placebo controlled study.

There are no simple clinical findings and specific laboratory changes that can be used to indicate the severity and progress of PPS. Different self-reporting questionnaires and objective measures of disability have often been used in clinical studies including SF-36 questionnaire, muscle strength measurement and walking test. The primary and secondary variables in this study were based on the clinical experience and literature reviewed.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects ≥18 to ≤75 years of age.
2. Post-polio syndrome according to Halstead and Gawne:

   * History of polio virus infection
   * Restitution or improvement regarding motor function and disabilities after initial infection
   * Confirmed polio by EMG
   * Subjectively increased muscular weakness after a period of at least 15 years functional stability
   * No other explanation but post-polio syndrome to the symptoms
3. Confirmed polio by EMG in the lower extremities in at least two of the following major muscle groups; musculi quadriceps, gastrocnemicus and tibialis anterior. (Two affected muscle groups in the same extremity were accepted).
4. Subjectively increased muscular difficulties or pain after a period of at least 15 years functional stability.
5. A muscle that had deteriorated within the last five years, and had 20-75 % of the muscle strength compared to age matched normal population when measured by a dynamometer or an electronic grip force sensor (GRIPPIT).
6. Stable weight (defined as weight change <7 kg) during the last five years.
7. Body Mass Index (BMI) £ 29 kg/m2.
8. Subjects capable to understand given information and had signed the Informed Consent Form after full discussion of the research nature of the treatment and its risks and benefits.

Exclusion Criteria:

1. Known or suspected intolerance to trial product or related products (e.g. sorbitol, glucose and fructose).
2. Selective IgA deficiency.
3. Inability to walk with walking aids.
4. Any active malignancy, history of active malignancy or treatment for malignancy during the last three years.
5. Disabling pain from extremities or skeletal system due to previous fracture(s), arthritis or other reasons not related to PPS.
6. Subjects who received or who within 12 weeks prior to enrolment received any immunosuppressive/ systemic corticosteroid treatment (topical corticosteroids excluded).
7. Treatment with intravenous human immunoglobulin for the Post-polio syndrome within six months prior to the first screening visit.
8. Participation in any other study during this study and the receipt of any investigational drug within three months prior to the screening visit.
9. Pregnancy or lactation or females of childbearing potential taking inadequate measures to prevent pregnancy.
10. Hepatitis or HIV disease.
11. Increased liver enzymes (ASAT, ALAT, γGT) above twice the upper normal value.
12. Creatine kinase >10 mkat/l.
13. Any disease or treatment that according to the discretion of the Investigator could pose a medical threat to the subject in combination with study drug, i.e. clinical manifested severe cardiovascular disease or severe arteriosclerosis or severe psychiatric disorder or other treatment that affected the immunological system such as prednisone and methotrexate.
14. Any disease or condition that according to the discretion of the Investigator would obstruct the subject from performing the tests in the protocol (e.g. fill in the questionnaires).
15. Conditions associated with a risk of poor protocol compliance (e.g. known drug or alcohol abuse).
16. Previous participation in the study.

Ages: 18 Years to 75 Years | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124
Dates: Start 2001-01; Study Completion 2003-05

PRIMARY OUTCOMES:
Primary endpoints:
Physical health was quantified using the SF-36 questionnaire scales summarized into the composite Physical Component Summary (PCS) measure.
Muscular strength was measured using a dynamometer or anelectronic grip force sensor (GRIPPIT) depending on the musclechosen.

SECONDARY OUTCOMES:
Secondary endpoints:
Functional balance was assessed by using the Timed "Up and Go" (TUG) test.
Activity pattern was assessed by the Physical Activity Scale of the Elderly (PASE).
Pain was assessed by a Visual Analogue Scale and by a pain drawing.
Fatigue was assessed using the Multidimensional Fatigue Inventory (MFI-20) questionnaire.
Vitality was assessed using the vitality subscale (VT) of SF-36 questionnaire.
Sleep was assessed using the Sleep quality scale.
Muscular strength measured by a dynamometer and an electronic grip force sensor (GRIPPIT) for those muscles not included as the primary endpoint.
Walking ability was assessed by a 6 minutes walking test.
Pulmonary capacity (vital capacity, FEV1, FEV %) was measured by a standard spirometer method.
Balance was assessed as postural sway velocity and the subject's ability to voluntarily sway to various locations in space (NeuroCom Balance Master) or balance assessed by static and dynamic posturography (Chattecx® balance system)
Adverse events
Vital signs (blood pressure and heart rate)
Physical examination
Laboratory tests

CONTACTS AND LOCATIONS:
Overall Officials: Kristian Borg, MD, Prof, Principal Investigator — Department of Rehabilitation Medicine;Huddinge University Hospital; Stockholm, Sweden
Locations (4):
- Sweden (4):
  - Danderyd Hospital, Danderyd
  - Sahlgrenska University Hospital, Gothenburg
  - Huddinge University Hospital, Stockholm
  - Uppsala Academic Hospital, Uppsala

REFERENCES:
- [Background] Gonzalez H, Khademi M, Andersson M, Wallstrom E, Borg K, Olsson T. Prior poliomyelitis-evidence of cytokine production in the central nervous system. J Neurol Sci. 2002 Dec 15;205(1):9-13. doi: 10.1016/s0022-510x(02)00316-7. PMID 12409177
- [Background] Gonzalez H, Khademi M, Andersson M, Piehl F, Wallstrom E, Borg K, Olsson T. Prior poliomyelitis-IVIg treatment reduces proinflammatory cytokine production. J Neuroimmunol. 2004 May;150(1-2):139-44. doi: 10.1016/j.jneuroim.2004.01.010. PMID 15081258
- [Result] Gonzalez H, Sunnerhagen KS, Sjoberg I, Kaponides G, Olsson T, Borg K. Intravenous immunoglobulin for post-polio syndrome: a randomised controlled trial. Lancet Neurol. 2006 Jun;5(6):493-500. doi: 10.1016/S1474-4422(06)70447-1. PMID 16713921
- See also: Pharmalink AB (sponsor) — http://www.pharmalink.se
- See also: PhD Disertation, Henrik Gonzalez, The post-polio syndrome: Studies of immunology and immunomodulatory intervention — http://diss.kib.ki.se/2005/91-7140-483-X/